CLINICAL TRIAL: NCT04144426
Title: Meal Schedule Effects on Circadian Energy Balance in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Terry Page, Professor Emeritus of Biological Sciences, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 140536
Record Dates: First submitted 2019-10-22; First posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Metabolism; Circadian Rhythms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal diet then modified diet (Experimental): Participates in the normal diet will receive 3 meals each day, breakfast at 8:00 AM,lunch at 12:30 PM and dinner at 5:45 PM. Participates in the modified diet skipped breakfast, had lunch at 12:30 PM, dinner at 5:45 PM, and a breakfast equivalent snack at 10:00 PM.
  Interventions: Behavioral: Normal diet; Behavioral: Modified diet
- Modified diet then normal diet. (Experimental): Participates in the modified diet skipped breakfast, had lunch at 12:30 PM, dinner at 5:45 PM, and a breakfast equivalent snack at 10:00 PM.Participates in the normal diet will receive 3 meals each day, breakfast at 8:00 AM,lunch at 12:30 PM and dinner at 5:45 PM.
  Interventions: Behavioral: Normal diet; Behavioral: Modified diet

INTERVENTIONS:
Behavioral: Normal diet — Participants will receive either a 2000 calorie or a 2500 calorie diet at normal meal times
Behavioral: Modified diet — Participants will receive either a 2000 calorie or a 2500 calorie diet with a single meal shift, breakfast is moved to an hour before bedtime.

SUMMARY:
This study will test will how eating on a particular daily schedule may effect energy, weight gain or loss, and body temperature.

DETAILED DESCRIPTION:
Although there have been a large number of studies in humans on the effects of food intake at night, very few studies directly address the hypothesis that inappropriately phased eating or snacking (i.e., at night) in humans disrupts metabolism and respiratory quotient (RQ) patterns and there are no studies that we are aware of that directly measure circadian clock phase relative to timing of food intake while evaluating metabolism. This may be critical, because it is well established that the timing of food intake can also modulate circadian clock phase.

Hypothesis: Food consumption in the subjective night (e.g., 20:00 - 02:00) will result in a different circadian metabolic profile measured by RQ) than food consumed in the subjective day.

Aim 1: To determine if there are daily rhythms of switching between lipid and carbohydrate metabolism in humans that are altered by the timing of food intake. Aim 2: To determine if timing of food intake results in "internal desynchronization" between the metabolic rhythms (RQ) and the rhythm in core body temperature (a marker of central circadian phase).

Aim 3: To determine if body composition has measurable impact on the circadian regulation of metabolism.

In this study we will test human subjects in a specially designed whole-room indirect calorimeter where energy expenditure and RQ will be monitored by indirect calorimetry continuously over 56 hours. Circadian phase and amplitude will be assessed by continuously recording the core body temperature rhythm using the Vital Sense Integrated Physiological Monitoring System in which subjects swallow a telemetry capsule that transmits core body temperature to a data acquisition module. In consultation with a nutritionist at Vanderbilt, we will use a cross-over design in which daily diets have the same caloric and nutritional value but in which the subjects consume the calories that would normally be breakfast as snacks consumed in the late-evening.

ELIGIBILITY:
Inclusion Criteria:

* Be able to understand the study, provide written informed consent (in English), and be able to fill out the questionnaire
* Be male or female older than 18 years of age;
* Have a normal BMI (20-25) or be obese (BMI more than 30);
* Have a normal basal glucose level (70-100 mg/dL)
* If female of childbearing potential, have a negative pregnancy test on study day;

Exclusion Criteria:

* Be pregnant or lactating;
* Have known sleep, metabolic (e.g., diabetes), or gastro-intestinal disorders except obesity;
* Had alcohol less than 24 hours before admission;
* Require assistance with activities of daily living;
* Have difficulty swallowing
* Be unable to complete a food and sleep diary
* Be smokers

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-10-08 (Actual); Primary Completion 2017-05-26 (Actual); Study Completion 2017-05-26 (Actual)

PRIMARY OUTCOMES:
Oxygen intake | 56 hours
  Subjects were housed in a whole room calorimeter and oxygen consumption was monitored minute by minute
Carbon dioxide exhaled | 56 hours
  Subjects were housed in a whole room calorimeter and carbon dioxide was monitored minute by minute
Core body temperature | 56 hours
  The subjects' circadian phase and amplitude will be assessed by continuously recording the core body temperature rhythm with an ingestible Vital Sense monitor.
Locomotor activity | 56 hours
  The subject's activity will be assessed throughout the experiment using a Actigraph (GT3X) triaxial monitor attached to the subject's wrist, waist, and ankle.

SECONDARY OUTCOMES:
Determination of Body Mass Index (BMI) | Baseline just prior to entry in the metabolic chamber
  A dual-energy X-ray absorptiometry (DXA) scan will be performed to assess subject's percentage body fat after check-in and before the first night in the metabolic chamber. Fat content will be used to accurately determine the subject's Body Mass Index.

CONTACTS AND LOCATIONS:
Overall Officials: Terry L Page, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No